CLINICAL TRIAL: NCT00554996
Title: Bacterial Interference for Prevention of Catheter-Associated UTI
Brief Title: Bacterial Interference for Prevention of Catheter-Associated UTI: Geriatric Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B4623-R
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Urinary Tract Infection
Keywords: urinary tract infection; urinary catheter; Escherichia coli; biofilm
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- E. coli 83972 coated urinary catheter (Other): E. coli 83972 coated urinary catheter
  Interventions: Device: E. coli 83972 coated urinary catheter

INTERVENTIONS:
Device: E. coli 83972 coated urinary catheter — E. coli 83972 coated urinary catheter

SUMMARY:
This study is a prospective pilot clinical trial investigating the use of urinary catheters coated with benign E. coli in geriatric subjects.

DETAILED DESCRIPTION:
1. Preparation of study catheters: Urinary catheters will be incubated in broth with E. coli 83972 for 48 hours prior to insertion into patients. Samples of broth will be removed after 24 hours and 48 hours of incubation to test for purity of the E. coli 83972. Study catheters will be inserted after 48 hours of incubation, unless contamination was seen on the 24-hour plates. The 48-hour plates will be read at 72 hours, and any contamination would prompt removal of the study catheter. For subjects who require antibiotics to clear their bladders prior to catheter insertion, we will use a derivative strain of E. coli 83972 with the appropriate antibiotic resistance.
2. Screening procedures: Eligible subjects will be identified by chart review and by discussion with health care providers. Research personnel will also periodically assess the inpatient geriatric beds and review upcoming appointments in the geriatric and urology clinics at the MEDVAMC. Potential outpatient subjects may be contacted by telephone before their clinic appointment to advise them of the study. Those wishing to participate will meet with study personnel in person when they come for their clinic appointment. At the time of enrollment, the principal investigator or the research coordinator will explain the study protocol in detail, and subjects will be given a chance to ask questions. Informed consent will be obtained from interested persons at that time. Any necessary screening procedures (history and physical examination, renal ultrasound, serum creatinine, baseline urine culture) will be performed after obtaining informed consent. Subjects who have not had a renal ultrasound within the past 12 months, or a serum creatinine measured within the past 6 months, will undergo these procedures. Also, study personnel will collect urine for culture to determine what organisms are present in the subject's bladder at baseline. The subject may receive 7-10 days of appropriate antibiotics to clear their bladders before insertion of study catheters, depending on the pre-existing bladder flora.
3. Insertion of study catheters: Subjects requiring fluoroquinolone antibiotics to clear their bladders will receive a study catheter 4-5 days after completing treatment. Subjects requiring any other class of antibiotics will receive a study catheter 2-3 days after completing antibiotic treatment. The study catheter will be inserted in by research personnel or by the unit nurse. Insertion will be performed using sterile technique. Urine will be collected through the newly inserted study catheters and cultured by study personnel.
4. Urine sample collection: Urine samples will be collected through the study catheter on days 1, 3, 7, 14, 21, and 28 after catheter insertion. Urine will be mailed to the PI's laboratory at the MEDVAMC in biological sample collection containers via overnight mail for outpatients, or the samples can be collected directly from inpatients.
5. Study catheter removal: A day 28 urine sample will be collected through the study catheter immediately prior to removal. Study catheters will be removed by study personnel at the MEDVAMC. Subjects who still have E. coli 83972 on the day of catheter removal will be given the option of taking antibiotics to eradicate the E. coli 83972 from the bladder or to remain colonized and in the follow-up phase of the study.
6. Specimen mailing procedure: We have utilized these specimen mailing supplies before. The study organism, E. coli 83972, has 83% survival after 72 hours in the specimen mailer tubes, when mailed from other locations in Texas and Louisiana. Both the study organism and other uropathogens have likewise been recovered from urinary catheters removed 72 hours previously and sent to us in specimen mailing tubes.
7. Microbiologic studies: Semi-quantitative cultures will be performed on each urine sample to determine whether E. coli 83972 is present and the relative concentration of each other species in the urine. The presence in the urine of bacteria other than E. coli will be examined using standard bacteriological methods only. E. coli strains will be assessed using standard microbiological techniques as well as molecular techniques in the research laboratory. Urine will be spread on MacConkey lactose agar plates and incubated to allow bacterial growth. Representative E. coli colonies will be subjected to restriction fragment length polymorphism (RFLP) analysis using pulse field gel electrophoresis (PFGE) to definitively identify E. coli 83972. The removed urinary catheters will be sonicated to extract surface-associated organisms. An aliquot of each sonicate will be plated for identification of organisms.
8. Defining outcomes: We will assess the safety and colonization success. For the purposes of this study, we will define successful bladder colonization as persistence of E. coli 83972 in the urine for > 28 days after insertion of the catheter. Shorter duration of colonization will be defined as failure to colonize the bladder. We will also compare the incidence of symptomatic UTI while colonized with E. coli 83972 to the incidence of symptomatic UTI experienced by the subjects in the year prior to study entry.
9. Safety assessment: The principal investigator will contact subjects daily for the first 3 days while they are wearing the study catheters, weekly for the remainder of the first 28 days after insertion of the study catheter, and monthly thereafter as long as they remain colonized with E. coli 83972. Subjects will be instructed to contact study personnel for signs or symptoms of UTI, catheter malfunction, or need for antibiotics.
10. UTI in elderly subjects can present with constitutional symptoms rather than those localized to the urinary tract, and the fever response can be blunted in the elderly. Symptomatic UTI will be defined as the presence of significant bacteriuria (>102 cfu/ml), pyuria (>10 WBC/hpf) plus > 1 of the following signs and symptoms: fever (> 100.0 F), suprapubic or flank discomfort, bladder spasm, malaise, altered functional status, or altered mental status, provided that no other etiologies for these clinical manifestations can be identified. Subjects' baseline incidence of UTI in the year prior to enrollment will be determined by chart review. Any documented treatment for UTI will be regarded as a symptomatic UTI. We will also inquire whether patients were treated for UTI at an outside facility. Subjects who develop symptomatic UTI will be treated with antibiotics guided by susceptibility patterns for the organism(s) grown from urine cultures.
11. Duration of participation: If a subject remains colonized with E. coli 83972 on day 28 after removal of the study catheter, and if the subject declines antibiotics to eradicate the study organism, we will continue to collect monthly urine specimens until the organism is lost from the bladder or until completion of 12 months, whichever comes first. Thus, an individual subject's participation in the study will be limited to 12 months or less.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed at the MEDVAMC
* Require an indwelling bladder catheter (either transurethral or suprapubic)
* Have a history of at least 1 UTI in the past will be eligible for enrollment
* Have pre-existing bladder colonization

Exclusion Criteria:

* obstructive urolithiasis
* percutaneous nephrostomy catheters
* supravesicular urinary diversion
* vesicoureteral reflux
* active malignancy
* uncontrolled diabetes mellitus
* AIDS
* requirement for immunosuppressive medication, expected survival < 6 months, creatinine clearance > 2.0 mg/dL, or current antibiotic therapy
* Latex allergy
* Allergic to 2 or more classes of drugs to which the urinary isolate is susceptible
* Prostate cancer on hormonal therapy with or without any surgery or radiation therapy anticipated within the next 6 months
* Prisoners
* Significant known mental illness or emotional disorder related to organic or inorganic causes
* subjects who are not capable of giving informed consent will not be included unless the subject's designated decision-maker is readily available

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Trautner, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

REFERENCES:
- [Background] Trautner BW, Cevallos ME, Li H, Riosa S, Hull RA, Hull SI, Tweardy DJ, Darouiche RO. Increased expression of type-1 fimbriae by nonpathogenic Escherichia coli 83972 results in an increased capacity for catheter adherence and bacterial interference. J Infect Dis. 2008 Sep 15;198(6):899-906. doi: 10.1086/591093. PMID 18643750
- [Background] Buscher A, Li L, Han XY, Trautner BW. Aortic valve endocarditis possibly caused by a Haematobacter-like species. J Clin Microbiol. 2010 Oct;48(10):3791-3. doi: 10.1128/JCM.00238-10. Epub 2010 Jul 7. PMID 20610676
- [Background] Desai DG, Liao KS, Cevallos ME, Trautner BW. Silver or nitrofurazone impregnation of urinary catheters has a minimal effect on uropathogen adherence. J Urol. 2010 Dec;184(6):2565-71. doi: 10.1016/j.juro.2010.07.036. PMID 21030042
- [Background] Qin G, Santos C, Zhang W, Li Y, Kumar A, Erasquin UJ, Liu K, Muradov P, Trautner BW, Cai C. Biofunctionalization on alkylated silicon substrate surfaces via "click" chemistry. J Am Chem Soc. 2010 Nov 24;132(46):16432-41. doi: 10.1021/ja1025497. Epub 2010 Oct 29. PMID 21033708
- [Background] Nelsen A, Trautner BW, Petersen NJ, Gupta S, Rodriguez-Barradas M, Giordano TP, Naik AD. Development and validation of a measure for intention to adhere to HIV treatment. AIDS Patient Care STDS. 2012 Jun;26(6):329-34. doi: 10.1089/apc.2011.0318. PMID 22680281
- [Background] Trautner BW, Gupta K. The advantages of second best: comment on "Lactobacilli vs antibiotics to prevent urinary tract infections". Arch Intern Med. 2012 May 14;172(9):712-4. doi: 10.1001/archinternmed.2012.1213. No abstract available. PMID 22782200
- [Background] Roig IL, Darouiche RO, Musher DM, Trautner BW. Device-related infective endocarditis, with special consideration of implanted intravascular and cardiac devices in a predominantly male population. Scand J Infect Dis. 2012 Oct;44(10):753-60. doi: 10.3109/00365548.2012.678882. Epub 2012 Jun 10. PMID 22681242
- [Background] Gupta K, Trautner B. In the clinic. Urinary tract infection. Ann Intern Med. 2012 Mar 6;156(5):ITC3-1-ITC3-15; quiz ITC3-16. doi: 10.7326/0003-4819-156-5-201203060-01003. No abstract available. PMID 22393148
- [Background] Trautner BW, Lopez AI, Kumar A, Siddiq DM, Liao KS, Li Y, Tweardy DJ, Cai C. Nanoscale surface modification favors benign biofilm formation and impedes adherence by pathogens. Nanomedicine. 2012 Apr;8(3):261-70. doi: 10.1016/j.nano.2011.11.014. Epub 2011 Dec 23. PMID 22197726
- [Background] Trautner BW, Hull RA, Thornby JI, Darouiche RO. Coating urinary catheters with an avirulent strain of Escherichia coli as a means to establish asymptomatic colonization. Infect Control Hosp Epidemiol. 2007 Jan;28(1):92-4. doi: 10.1086/510872. Epub 2006 Dec 29. PMID 17230395
- [Background] Trautner BW, Hull RA, Darouiche RO. Escherichia coli 83972 inhibits catheter adherence by a broad spectrum of uropathogens. Urology. 2003 May;61(5):1059-62. doi: 10.1016/s0090-4295(02)02555-4. PMID 12736047
- [Background] Nelsen A, Gupta S, Trautner BW, Petersen NJ, Garza A, Giordano TP, Naik AD, Rodriguez-Barradas MC. Intention to adhere to HIV treatment: a patient-centred predictor of antiretroviral adherence. HIV Med. 2013 Sep;14(8):472-80. doi: 10.1111/hiv.12032. Epub 2013 Apr 3. PMID 23551395
- [Background] Marschall J, Carpenter CR, Fowler S, Trautner BW; CDC Prevention Epicenters Program. Antibiotic prophylaxis for urinary tract infections after removal of urinary catheter: meta-analysis. BMJ. 2013 Jun 11;346:f3147. doi: 10.1136/bmj.f3147. PMID 23757735
- [Background] Trautner BW, Petersen NJ, Hysong SJ, Horwitz D, Kelly PA, Naik AD. Overtreatment of asymptomatic bacteriuria: identifying provider barriers to evidence-based care. Am J Infect Control. 2014 Jun;42(6):653-8. doi: 10.1016/j.ajic.2014.02.003. Epub 2014 Apr 6. PMID 24713596
- [Result] Horwitz D, McCue T, Mapes AC, Ajami NJ, Petrosino JF, Ramig RF, Trautner BW. Decreased microbiota diversity associated with urinary tract infection in a trial of bacterial interference. J Infect. 2015 Sep;71(3):358-367. doi: 10.1016/j.jinf.2015.05.014. Epub 2015 Jun 3. PMID 26048203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E. Coli 83972 Coated Urinary Catheter
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: See Eligibility section.
Arm/Group | E. Coli 83972 Coated Urinary Catheter
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 70.9 [58 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Rate of UTI While Colonized With E. Coli 83972.
Description: Rate of UTI during colonization with E. coli 83972.
Time Frame: 0-266 days of colonization
Population: Number of UTIs per 1000 patient-days during colonization with E. coli 83972.
Measure: Number; unit: UTIs per 1000 patient-days
Arm/Group | E. Coli 83972 Coated Urinary Catheter
Number analyzed (Participants) | 10
UTIs per 1000 patient-days | 8.5

ADVERSE EVENTS:
Arm/Group | E. Coli 83972 Coated Urinary Catheter
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E. Coli 83972 Coated Urinary Catheter (N=10)
Febrile UTI or Urosepsis/bacteremia (Renal and urinary disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Our trial was a small study with no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes